CLINICAL TRIAL: NCT01274078
Title: Effects of Exercise With or Without Blueberries on Cardiovascular Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, MD professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FHN_exc_blueberries
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Risk Factors Cardiovascular Disease; Inflammation; Exercise; Sedentary Life
Keywords: inflammation; lipids; CRP
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — blueberry extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional food (No Intervention): Regular eating habits during exercise period
- Blueberries (Active Comparator): Intervention: Addition of blueberries (150g/day) to regular food during the exercise period on days with exercise
  Interventions: Biological: Blueberries

INTERVENTIONS:
Biological: Blueberries — 150 grams of frozen blueberries on the same day as exercise
  Arms: Blueberries

SUMMARY:
About 32 healthy subjects are subjected to 4 weeks of exercise, 4 weeks of washout and 4 weeks of sedentary life style, randomization decides whether they start with exercise or with being "couch potatoes". All participants are also randomized to also consume 150 g of blueberries on exercise days or not. The exercise is constituted of 5 km running 5 days a week during the 4 week period. The exercise period and the "couch" period are started and ended with a 5 km run at maximal speed and the fasting blood samples for cardiovascular risk factors are measured before and after this run, ie 8 times in total.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* significant disease and disabilities that hinder running

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
markers for cardiovascular disease | 3 months
  Insulin levels, glucose levels, lipids, hs-CRP, troponin T

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping, Sweden